CLINICAL TRIAL: NCT01789151
Title: 99mTc-labelled D-Glucosamine in the Evaluation of Disease Activity in Patients With Degenerative and Inflammatory Rheumatic Conditions
Brief Title: 99m-Technetium- Glucosamine in Arthritis
Status: No longer available | Type: Expanded Access
Sponsor: University of Sydney (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: Glucosamine; IMM 11-0091 (Other: WSLHD HREC)
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis
Keywords: arthritis; nuclear imaging; rheumatoid; ankylosing spondylitis; glucosamine
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis

INTERVENTIONS:
Device: Technetium labelled glucosamine — Nuclear medicine imaging of arthritic joints using radioactive glucosamine

SUMMARY:
Preliminary data following a pilot study from our institution confirms the ability of 99mTc-glucosamine (99mTc-ECDG) to differentiate between active, subclinical and quiescent disease in patients with rheumatoid arthritis, scleroderma lung, and vasculitis. We propose to extend these findings and further evaluate this imaging modality for its clinical utility, limitations, and application.

An unacceptably high level of morbidity exists amongst patients suffering from rheumatic disease. This is often the result of mild disease being missed or misdiagnosed, and therapy inordinately delayed or inappropriate. The currently used therapeutic agents themselves have associated side-effects adding to unfavourable clinical outcomes. There is therefore a need for a superior, less expensive and more easily accessible imaging modality to assess the degree of inflammation to guide the clinician. Glucosamine is absorbed and metabolised in a manner not too dissimilar to that of glucose, and it can be readily labelled to form 99mTc-ECDG. Scans can be acquired within 3 hours of intravenous administration of this agent, accurately depicting sites of active inflammation/disease.

HYPOTHESIS Glucose is a vital cellular substrate that accumulates at inflamed tissues because of the greater metabolic needs of the cells during active disease. Glucosamine, being an analogue of glucose, is metabolised more quickly in inflamed than non-inflamed tissue and thus 99mTc-ECDG scintigraphy like 18-Fluorodeoxyglucose (18FDG-PET) scintigraphy allows for detection of active inflammation. Unlike current bone scans this agent has the sensitivity to detect subclinical inflammatory disease that would in turn provide essential information to ensure accurate diagnosis and treatment.

DETAILED DESCRIPTION:
Aim 1. To evaluate the role of 99mTc-ECDG in Rheumatoid Arthritis (RA). Both as a monitoring and diagnostic tool.

Approach. Three separate cohorts of patients suffering from RA will be recruited;

1. Patients with newly diagnosed RA;
2. Patients with active and long-standing RA before and after treatment with anti-TNF;
3. Patients with RA in remission with or without anti-TNF treatment.

5-10 patients will be recruited into each cohort. In order to provide written consent all patients will be older than 18 years old. Exclusion criteria will include any patient with an allergy to glucosamine or seafood, any patient with end-stage renal or hepatic disease, pregnancy or lactation. No restrictions will be imposed on the treatment patients are able to receive for their underlying rheumatic condition, nor for any other medical condition while in this study. Patients will be required to cease any glucosamine therapy for three days prior to the injection of the radiotracer.

An evaluation of patient's history and physical examination will be conducted prior to tracer administration. All relevant disease will be documented as well as concurrent illnesses and treatment regimes. A rheumatologist will assess disease severity and documented as per recommendations outlined under the PBS guidelines for subsidised treatment (HIC - Medicare Australia). Biological markers of disease will be acquired from each patient at the time of clinical assessment, including ESR, CRP levels, rheumatoid factor and anti-citrullinated peptide antibodies. Similar assessments will be undertaken at six monthly intervals for three years. These results will be used to correlate with the scan findings. Patients from cohort A & B will have their initial scans acquired prior to the commencement of therapy. Scans will be repeated six months later in all patients. Results will be analysed on both a per patient basis and a per joint basis.

AIM 1a. To correlate 99mTc-ECDG joint uptake with clinical parameters of disease.

The scan findings of each group will be graded by a nuclear medicine physician (SA) noting the pattern of tracer uptake and the intensity of tracer uptake. Relative tracer activity in joints will be correlated with the activity in the brain / skull (where essentially no uptake is evident). In addition, the neighbouring muscle tissue, the liver and the cardiac blood pool activity at the two scanning time points (15 and 120 minutes) will be evaluated. A four point (0-3) grading system will be utilised to semi-quantify the scan findings, and is as follows:

0 - Nil uptake - defined as no increased / minimally increased tracer activity in region of interest (ROI; activity approximates uptake in the brain);

1. - Mild - tracer uptake in ROI approximates that of the neighbouring muscle tissue;
2. - Moderate - tracer uptake in ROI is greater than that in the vicinity of the heart; and,
3. - Severe - tracer uptake in ROI approximates that of the liver. The scan findings will then be compared to clinical parameters as documented at the time of the study and on follow-up assessment (as outlined under aim 1). This will enable the investigators to assess disease progression or remission over time. It will thus be possible to evaluate the predictive nature of the scan findings in this respect.

AIM 1b. To evaluate 99mTc-ECDG joint uptake differences before and after treatment. That is, to predict response to therapy. One of the purposes of follow-up is to identify changes in disease activity over time. The clinical and scan findings at the time of recruitment will be compared to the corresponding findings from the follow-up assessments (as outlined in Aim 1 & 1a). Patients from cohorts A & B will permit assessment of clinical response to therapy. Thus, any regression of disease activity or otherwise, can be correlated with the differences as depicted on the scans acquired at baseline and at six months later. In cohort B, the 99mTc-ECDG scans acquired at baseline and 6 months later from inadequate responders to conventional therapy will be compared to those with a favourable clinical response.

Follow-up studies in patients from cohort C (disease in remission) will provide information regarding:

* the reproducibility of the scan findings in patients who remain clinically stable,
* the significance of probable subclinical disease (increased tracer uptake in joints of patients who are otherwise asymptomatic on the baseline study and the changes observed on the follow-up scans),
* and the sensitivity in detecting recurrent disease (changes in tracer distribution in joints that become inflamed in the intervening period).

AIM 1c. To correlate between findings on 99mTc-ECDG with other imaging modalities, including bone scintigraphy and 18FDG-PET scintigraphy. In at least 3 RA patients with a wide range of disease activity, a bone scan will be performed within 72h of the 99mTc-ECDG. At least 3 patients will also undergo 18FDG-PET scintigraphy. These scans will be evaluated by an experienced nuclear medicine physician (SA), and correlated to the patient profile and the 99mTc-ECDG scan findings. These cohorts will enable the value of the different clinical information provided by each imaging technique and their complementary nature to be evaluated. It is anticipated that this study will take 30 months to complete. All patients will be recruited with the aim to recruit all patients in the first 12 months and followed up for at least 24 months.

AIM 2. To investigate the role of 99mTc-ECDG in detecting seronegative spondyloarthritis. Distinguishing back-pain related to disease flare-up/progression and alternative causes (osteoarthritis, disc pathology) in patients with early AS is difficult. Therapy is cause-specific. Inappropriate application of therapeutic regimes can delay recovery often leading to unforeseen complications with poor outcomes (eg. steroid-related osteoporotic vertebral crush fractures). Plain X-rays, CT scans and MRI will effectively highlight the irreversible chronic changes of this disease. However, these techniques seldom detect the earliest pathogenic changes, being the most amendable to therapeutic intervention. 99mTc-ECDG, by virtue of its ability to accumulate at sites of inflammation, appears successful in identifying early and mild disease. Furthermore, the pattern of tracer distribution will assist in differentiating between the competing diagnoses. A control group of 10-15 patients with mechanical back pain will be used as controls 10-15 AS patients with varying degrees of disease activity will be recruited. TNF-alpha inhibitor therapy will be administered to patients meeting the necessary guidelines and scans performed pre and post treatment. Repeat studies will be acquired 6 months later in all patients. A comparison of clinical findings, documented by experienced Rheumatologists with regular six-monthly follow-up over three years will be conducted. The predictive value of these scans with respect to treatment response will also be assessed as outlined in Aim 1b. MRI scans, the gold standard for sacro-ileitis, will be acquired within 72 hours of the 99mTc-ECDG scans, for comparison of findings in the lumbo-sacral region. A number of these patients will also undergo bone scintigraphy and / or 18FDG-PET scintigraphy (as outlined in Aim 1c), to evaluate the comparative value of these alternate imaging modalities.

ELIGIBILITY:
Inclusion Criteria:

* In order to provide written consent all patients will be older than 18 years old. Patients with RA need to satisfy the ACR criteria. Similarly for AS patients need to satisfy current criteria for the diagnosis.

Exclusion Criteria:

* Exclusion criteria will include any patient with an allergy to glucosamine or seafood, any patient with end-stage renal or hepatic disease, pregnancy or lactation. Patients with previous history of malignancy, TB, Hep B, Hep C, AIDS will be excluded.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Manolios, MD, Phd, Principal Investigator — University of Sydney / Westmead Hospital; Nicholas Manolios, Principal Investigator — University of Sydney / Westmead Hospital
Locations (1):
- Westmead Hospital, Sydney, New South Wales, Australia